CLINICAL TRIAL: NCT06262334
Title: Developing a Community-Informed, Peer-to-Peer Intervention to Improve Health-Related Quality of Life Among African American Men
Brief Title: Evaluating the Fade to Fitness Program: A Barbershop-based Program for Black Men
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Guillermo Wippold, Associate Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00133917; K23MD016123 (NIH)
Record Dates: First submitted 2024-01-17; First posted 2024-02-16 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-03

CONDITIONS: Health Related Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The Fade to Fitness Program (Experimental)
  Interventions: Behavioral: The Fade to Fitness Program

INTERVENTIONS:
Behavioral: The Fade to Fitness Program — The Fade to Fitness Program is a group-based and barbershop-based behavioral intervention to improve health-related quality of life among African American men. The program is unique because it is culturally targeted and individually tailored. The culturally targeted content was developed following barbershop-based focus groups. The Fade to Fitness Program targets four behaviors strongly linked to health-related quality of life among African American men - physical activity, healthy eating, stress management, and depression management. During the group-based portion of the program, Motivational Interviewing is used by the facilitator as a conversational approach to enhance participants' motivation and commitment towards positive behavior change. The goal is to foster intrinsic motivation among participants to engage in these behaviors. It is individually tailored by encouraging participants to identify personal values and linking them to health promoting behaviors.

SUMMARY:
The Fade to Fitness Program is a targeted intervention designed to improve the holistic health and quality of life among Black men. This comprehensive initiative focuses on four key health behaviors: Physical Activity, Healthy Eating, Stress Management, and Depression Management.

It is grounded in psychological and social theories like Self-Determination Theory, Motivational Interviewing, and Social Cognitive Theory. The program emphasizes the importance of making informed choices, feeling competent and connected, and learning through observation and modeling. Facilitators play a pivotal role, leading group discussions, providing support, and fostering an inclusive atmosphere.

The program is structured into weekly sessions that tackle each health behavior, interspersed with off weeks; for community engagement, especially in barbershops, to discuss health topics and promote a healthier lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American or Black American male - 18 - 90 years of age
* Able to speak and understand English

Exclusion Criteria:

* Currently participating in another health promotion intervention
* On a special diet for a serious health condition
* Intending to move within 6 months of participating in the intervention

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals must identify as male regardless of biological sex.
Enrollment: 15 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of men who are eligible/eligible. | Up to 1 week
  An excel sheet will be used to track the number of men who express interest in the study and are eligible/ineligible.
Length of time needed to enroll 15 men | Up to 1 week
  An excel sheet will be used to track length of time needed to enroll 15 men.
Facilitator-assessed attendance in intervention | Up to 1 week
  An excel sheet will be used to track each participant's attendance. Participants attendance will be entered as 1 (attended) or 0 (did not attend).
Number of men who express interest in the study | Up to 1 week
Attrition in intervention | Baseline to 5 months
  The excel sheet used to assess attendance will be used to assess attrition.
Acceptability, appropriateness, demand, implementation, practicality, and integration of the intervention | 2 months
  Qualitative data will be collected based on guidelines created by research funded by the National Cancer Institute to understand the feasibility of health promotion interventions among underserved populations. The interview questions will assess the acceptability (e.g., satisfaction, perceived appropriateness, fit with cultural structure), demand (e.g., intent to use, actual use, expressed interest or intention to use), implementation (e.g., degree of execution), practicality (e.g., amount of time needed, quality of implementation, ability to carry out intervention activities), and integration (e.g., perceived sustainability) of the intervention.

SECONDARY OUTCOMES:
Change in weight | Change from baseline to 5 months
Change in body mass index | Change from baseline to 5 months
Change in moderate-to-vigorous physical activity | Baseline to 5 months
  Average minutes of moderate-to-vigorous physical activity measured over 5 consecutive days using an accelerometer
Global Health - Mental 2a | Baseline to 5 months
  2-item measure of mental health; range: 2 - 10 with higher scores indicating better mental health.
Global Health - Physical 2a | Baseline to 5 months
  2-item measure of physical health; range: 2 - 10 with higher scores indicating better physical health.
Perceived Stress Scale | Baseline to 5 months
  10-item measure of perceived stress; range: 0 - 40 with higher scores indicating more perceived stress.
Emotional Distress - Depression - Short Form 4a | Baseline to 5 months
  4-item measure of depression; range: 4 - 20 with higher scores indicating more depressive symptoms.
Healthy Eating Subscale of the Health Promotion Lifestyle Profile II | Baseline to 5 months
  9-item measure of healthy eating; range: 9 - 36 with higher scores indicating greater engagement in healthy eating.
Instrumental Support- Short Form 4a | Baseline to 5 months
  4-item measure of instrumental support; range: 4 - 20 with higher scores indicating more instrumental support.
Informational Support - Short Form 4a | Baseline to 5 months
  4-item measure of informational support; range: 4 - 20 with higher scores indicating more informational support.
Emotional Support - Short Form 4a | Baseline to 5 months
  4-item measure of emotional support; range: 4 - 20 with higher scores indicating more emotional support.
Companionship - Short Form 4a | Baseline to 5 months
  4-item measure of companionship; range: 4 - 20 with higher scores indicating more companionship.
Motivation and Attitudes Towards Changing Health (MATCH) | Baseline to 5 months
  9-item measure of health motivation; range: 9 - 45 with higher scores indicating greater health motivation.
NIH Self-Efficacy Measure | Baseline to 5 months
  10-item measure of health self-efficacy; range: 10 - 50 with higher scores indicating greater health self-efficacy.
Subjective Social Norms of Health Behavior | Baseline to 5 months
  4-item measure using a researcher-developed subjective social norms measure to engage in health behaviors; range: 4 - 28 with higher scores indicating fewer social norms to engage in health behaviors.
Valuing Questionnaire | Baseline to 5 months
  10-item measure to assess values-based behavior; range: 0 - 60 with higher scores indicating more values-based behaviors.
Diet | Baseline to 5 months
  Measure using the Dietary Screener Questionnaire (variable length). This measure assess amount of dietary intake of fruits, vegetables, fiber, added sugars, calcium, dairy, and whole grains. A higher response indicates more intake of fruits, vegetables, fiber, added sugars, calcium, dairy, and whole grains.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo M Wippold, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared upon reasonable request.
URL: https://www.sc.edu